CLINICAL TRIAL: NCT04060212
Title: Microbial Mechanisms of Methylmercury Metabolism in Humans
Brief Title: Mercury Metabolism by Bacteria in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Matthew Rand, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3842; R01ES030940 (NIH)
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Mercury--Toxicology
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): All participant will eat 6 meals of tuna fish. All participants will take a prebiotic dietary supplement.
  Interventions: Other: Tuna fish; Dietary Supplement: prebiotic

INTERVENTIONS:
Other: Tuna fish — Six meals of tunafish (~200gms) will be consumed. Three meals will be consumed in a period of 14 days, and a subsequent 3 meals will be consumed within a 14 day period six month after the first 3 meals.
Dietary Supplement: prebiotic — Prebiotin brand prebiotic will be consumed at 8grms/day for a period of 75 days. The prebiotic administration will begin with the second grouping of 3 fish meals.

SUMMARY:
The purpose of this study is to evaluate how the bacteria in your gut can improve the break-down and de-toxification of non-harmful levels of a naturally occurring form of mercury (methylmercury) that comes with eating fish. This research could help scientists and doctors understand whether or not mercury in fish that we are likely to eat poses any concern for the health of people.

DETAILED DESCRIPTION:
The overall objective of this study is to investigate the role of gut microbes in mediating how humans metabolize and excrete the environmental neurotoxicant methylmercury (MeHg). Exposure to MeHg through consumption of fish continues to pose a health risk for many populations globally. There remains considerable uncertainty in advising the public on mercury risks associated with fish consumption. A great deal of uncertainty stems from the fact that the MeHg metabolism and elimination rate is known to vary widely from individual to individual. This translates into the possibility that two individuals consuming the same amount of fish with the same frequency could, unknowingly, experience as much as 4-fold difference in accumulation of MeHg in their bodies. Thus, there is a need for greater understanding of the mechanisms of MeHg metabolism and elimination, as well as for development of tools to assess these characteristics in people. Our scientific premise is that symbiotic microbes in the human gut are required for the efficient biotransformation (demethylation) and excretion of toxic MeHg. In this prospective intervention study we will examine the variation in the rate at which MeHg is excreted, both between human subjects and within subjects over time, and relate it to the MeHg demethylation activity that is harbored in their respective gut microbes. Furthermore, through intervention with a prebiotic dietary supplement, we will induce a change in the gut microbial composition within the same individual and evaluate if slower of faster MeHg metabolism ensues. With these approaches we will obtain gut microbiome samples that correlate with faster or slower MeHg elimination kinetics. We then aim to identify specific genera and species of bacteria in the human gut responsible for MeHg metabolism. We will do this by feeding volunteers fish meals with documented trace levels of MeHg that are below any harmful level of exposure. We will subsequently measure kinetic rates of MeHg elimination via mass-spectrometry analysis of hair strands. We will also sample feces from the subjects as a source of the gut microbiota and as a medium to analyze the extent of MeHg metabolism (demethylation) that parallels its elimination. Study team members at Montana State University will directly examine the ability of the human gut microbiota to induce MeHg metabolizing activity in germ-free mice at rates that correspond with that seen in the human subject it was derived from. In parallel, we will use metagenomic sequence-informed strategies to bring isolated strains of the human gut bacteria to culture and subsequently interrogate their MeHg demethylating activity. We anticipate our results will lead to a clearer understanding of the microbial basis of human MeHg metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18-80 years in age.
* Subjects must be in good general health based on self-reported health status, with the exception of self-reported conditions listed in the exclusion criteria.
* Subject must be willing to comply with study procedures.

Exclusion Criteria:

* Known allergy to fish.
* Pregnant or lactating women.
* Use of hair dyes or chemical treatments within the prior month and/or intent to use such treatments during the two trial periods. (Hair treatment during the washout period up to one month prior to the second trial is acceptable).
* Known gastrointestinal or renal disorders.
* Subjects with diminished mental capacity.
* Use of antibiotics within two months leading up to the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Coe GL, Krout IN, Munro-Ehrlich M, Beamish CR, Vorojeikina D, Colman DR, Boyd EJ, Walk ST, Rand MD. Assessing the role of the gut microbiome in methylmercury demethylation and elimination in humans and gnotobiotic mice. Arch Toxicol. 2023 Sep;97(9):2399-2418. doi: 10.1007/s00204-023-03548-7. Epub 2023 Jul 1. PMID 37392210

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 36
Completed | 29
Not Completed | 7
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: years] | 32.6 [23 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Mercury Elimination Rate Before Pre-biotic
Description: Mercury elimination rate will be determined for each individual at the beginning of the study, prior to any prebiotic administration. This determination will take place over the first 75 days of the study, wherein the first three fish meals are consumed, a eliminaiton period follows and then hair is sampled and analyzed. Time-resolved levels of mercury will be determined by longitudinal analysis of single hair strands using mass spectrometry methods. The values will be used to calculate the mercury elimination rate for each individual. The average elimination rate across the cohort before prebiotic will be reported. This total analysis will require approximately 2.5 months.
Time Frame: 2.5 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 29
days | 48.5 (14.5)

2. Primary Outcome: Mercury Elimination Rate After Pre-biotic
Description: Mercury elimination rate will be determined for each individual after commencing prebiotic self-administration for a period of 75 days, contemporaneously with the second set of fish meal consumption. This will begin approximately 6 months after the finish of the first round of fish meals and elimination (i.e. approximately 8.5 months after the participant starts the study). This second round will last approximately 2.5 months. Time-resolved levels of mercury will be determined by longitudinal analysis of single hair strands using mass spectrometry methods. The values will be used to calculate the mercury elimination rate for each individual. The average elimination rate across the cohort after prebiotic, from approximately 8.5 to 11 months will be reported.
Time Frame: 11 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 29
days | 49.1 (14.3)

3. Secondary Outcome: Change in Mercury Metabolism Ratio
Description: Mercury metabolism ratio, i.e. conversion of methylmercury to inorganic mercury, will be determined for each individual before and after prebiotic administration. The difference in average metabolism ratio across the cohort before and after prebiotic will be reported. Mercury elimination ratios will be measured in stool samples using mass spectrometry methods.
Time Frame: Baseline to 10 months
Population: This data was not collected because a flaw was discovered in the analytical design.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 3/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=36)
nausea (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT04060212/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT04060212/ICF_001.pdf